CLINICAL TRIAL: NCT05533021
Title: Impact of the Training Structured According to Meleis's Transition Theory on Postpartum Difficulties and Quality of Life in Primipara Mothers
Brief Title: Meleis's Transition Theory on Postpartum Difficulties and Quality of Life in Primipara Mothers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Collaborators: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Ayla KORKMAZ, Assistant Professor, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-KAEK-033
Record Dates: First submitted 2022-09-01; First posted 2022-09-08 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Postpartum Care; First Birth; Cesarean Section
Keywords: Depression; Difficulty; Meleis's Transition Theory; Postpartum Period; Primipara Mother; Quality of Life
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: randomized controlled experimental study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Training and consultancy
  Interventions: Other: Training and Consultancy
- control group (No Intervention): Standard postpartum care

INTERVENTIONS:
Other: Training and Consultancy — In order to facilitate the transition to motherhood, theory-based training and counseling was provided to primiparous mothers on self and infant care.
  Arms: intervention group

SUMMARY:
The randomized controlled experimental study sought to determine the impact of the training structured according to Meleis's Transition Theory on postpartum difficulties and quality of life in primipara mothers.

DETAILED DESCRIPTION:
In the study, the intervention group (39 mothers) was given face-to-face training in the hospital, which was structured according to Meleis' Transition theory, 24 hours after the cesarean section.Telephone counseling was provided on the 5th, 15th and 42nd days after discharge. Thus, these mothers were followed up 4 times in the postpartum period. No intervention was made in the control group (40 mothers).

ELIGIBILITY:
Inclusion Criteria: Mothers with the following criteria were included in the study;

* Primiparous
* Cesarean delivery
* Over 18 years old
* At least primary school graduate
* Communicating verbally
* Using mobile phone and whatsapp application
* Married and living with spouse

Exclusion Criteria: Mothers with the following criteria were excluded from the study;

* Having a risky pregnancy history
* Having a history of chronic disease
* Diagnosed with a psychiatric illness
* Having a health problem in herself or her baby that requires separation from each other
* Having a baby with any congenital anomaly or severe disease detected at birth

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — focused on postpartum mothers
Enrollment: 79 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2022-01-28 (Actual)

PRIMARY OUTCOMES:
Change in the level of difficulty in self-care of primipara mothers in post-cesarean (42 days) | 1st follow-up (pre-training), 2nd follow-up (post-cesarean 5th day), 3rd follow-up (post-cesarean 15th day) and 4th follow-up (post-cesarean 42nd day)
  Change in the level of difficulty in self-care of primipara mothers in post-cesarean (42 days) was evaluated with a form prepared by the researchers using the literature. This form consists of 15 Likert type items. Each item is scored between 0 and 2. Therefore, the minimum score of the form is 0, while the maximum score of the form is 30. If the score obtained from the form is high, the difficulty level is high, and if the score obtained from the form is low, the level of difficulty is low.
Change in the level of difficulty in baby-care of primipara mothers in post-cesarean (42 days) | 1st follow-up (pre-training), 2nd follow-up (post-cesarean 5th day), 3rd follow-up (postcesarean 15th day) and 4th follow-up (postcesarean 42nd day)
  Change in the level of difficulty in baby-care of primipara mothers in post-cesarean (42 days) was evaluated with a form prepared by the researchers using the literature. This form consists of 9 Likert type items. Each item is scored between 0 and 2. Therefore, the minimum score of the form is 0, while the maximum score of the form is 18. If the score obtained from the form is high, the difficulty level is high, and if the score obtained from the form is low, the level of difficulty is low.
Postpartum depression | Post-cesarean 42nd day
  Edinburgh postpartum depression scale consists of 10 questions. The answers are evaluated in a 4-point Likert format and scored between 0-3. The total score of the scale is obtained by summing these item scores. Persons with a score above 12 points are considered a risk group. The lowest score is 0 and the highest score is 30.
  Primiparous mothers filled out the google form via whatsapp at the first interview (pre-training) and post-cesarean the 42nd day
Postpartum quality of life | Post-cesarean 42nd day
  Postpartum quality of life scale is a likert-type scale consisting of five sub-dimensions and a total of 40 items. Each item is evaluated for its importance and satisfaction for the mother. The Quality of Life Score is in the range of 0-30. Primiparous mothers filled out the google form via whatsapp at the first interview (pre-training) and post-cesarean the 42nd day

CONTACTS AND LOCATIONS:
Overall Officials: Ayla KORKMAZ, Asst.Prof., Principal Investigator — Tokat Gaziosmanpasa University
Locations (1):
- Tokat Gaziosmanpaşa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No